CLINICAL TRIAL: NCT00555945
Title: Re-Evaluation of GAmma3 Intramedullary Nails in Hip Fracture: A Multi-Centre Randomized Controlled Trial of Gamma3 Intramedullary Nails Versus Sliding Hip Screws in the Management of Intertrochanteric Fractures of the Hip
Brief Title: Re-Evaluation of GAmma3 Intramedullary Nails in Hip Fracture (REGAIN)
Acronym: REGAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stryker Trauma and Extremities (Industry)
Collaborators: Stryker Osteosynthesis (Unknown); Global Research Solutions (Industry)
Responsible Party: Nils Reimers, Stryker Trauma GmbH
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 06042011_REGAIN_v1.0
Record Dates: First submitted 2007-11-07; First posted 2007-11-09 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2011-06

CONDITIONS: Femoral Neck Fractures; Intertrochanteric Fracture
Keywords: Intertrochanteric fracture; Gamma3 intramedullary nail; Sliding hip screw
MeSH Terms: conditions — Femoral Neck Fractures; Hip Fractures | interventions — Fracture Fixation, Intramedullary

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Gamma3 intramedullary nail
  Interventions: Procedure: Gamma3 intramedullary nail (Stryker)
- 2 (Active Comparator): Sliding hip screw
  Interventions: Procedure: Sliding Hip Screw

INTERVENTIONS:
Procedure: Gamma3 intramedullary nail (Stryker) — The Gamma3 nail is cannulated for Guide-Wire-controlled insertion, and features a conical tip for optimal alignment with the inner part of the cortical bone. A single distal Locking Screw is provided to stabilize the nail in the medullary canal and to help to prevent rotation in complex fractures.
  Other Names: Gamma Nail; Gamma3 Nail; Intramedullary Nail (IM Nail)
  Arms: 1
Procedure: Sliding Hip Screw — The sliding hip screw is a single larger diameter partially threaded screw, which is affixed to the proximal femur with a side plate (with a minimum of two holes and a maximum of four holes) and no supplemental fixation.
  Other Names: Sliding Hip Screw (SHS); Dynamic Hip Screw (DHS); Compression Screw and Side Plate
  Arms: 2

SUMMARY:
The purpose of this study is to assess the impact of Gamma3 intramedullary nails versus sliding hip screws on rate of revision surgery in individuals with inter-trochanteric fractures. Secondary outcomes include fracture healing rates, fracture related complications, and health-related quality of life.

DETAILED DESCRIPTION:
Hip fractures are becoming a more prevalent issue worldwide, leading to profound morbidity, and in some cases, mortality. Currently the most common method of surgical treatment includes the use of a sliding hip screw over a Gamma intramedullary nail, but there is conflicting evidence regarding which device has a lower revision of surgery rate and complication rate. The newest generation of Gamma3 nails have strong rationale suggesting significantly decreased rates of femoral shaft fractures and improved function. The improvements in implant design of the Gamma3 nail provide compelling rationale for the conduct of a large, definitive trial, and therefore a pilot study is being conducted to confirm or refute our ability to recruit patients and assess the consistency between site estimates and actual recruitment, determine the degree to which site investigators can adhere to trial protocol, confirm or refute our anticipated ability to achieve close to 100% follow- up, assess our ability to maintain 100% data quality, field test our case report forms for clarity and appropriateness, and to determine whether we can successfully manage the logistics of coordinating trial activities across multiple sites.

This trial is a pilot, multi-center, concealed randomized controlled trial. Surgeons will use one of the two surgical strategies in patients who have sustained a trochanteric fracture; the Gamma3 intramedullary nail or the sliding hip screw. Clinical assessments will occur at the time of hospital admission, 1 week, 3 months, 6 months, and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Adult men or women aged 50 years and older (with no upper age limit).
* An trochanteric fracture (stable or unstable) confirmed with anterior and posterior lateral hip radiographs, computed tomography, or magnetic resonance imaging (MRI).
* Operative treatment within 3 days (i.e., 72 hours) after the trauma.
* Patient was ambulatory prior to fracture, though they may have used an aid such as a cane or a walker.
* Anticipated medical optimization of the patient for operative fixation of the proximal femur.
* Provision of informed consent by patient or proxy.
* Low energy fracture (defined as a fall from standing height).
* No other major trauma.

Exclusion Criteria:

* Associated major injuries of the lower extremity (i.e., ipsilateral or contralateral fractures of the foot, ankle, tibia, fibula, knee, or femur; dislocations of the ankle, knee, or hip; or femoral head defects or fracture).
* Retained hardware around the affected hip.
* Infection around the hip (i.e., soft tissue or bone).
* Patients with disorders of bone metabolism other than osteoporosis (i.e., Paget's disease, renal osteodystrophy, or osteomalacia).
* Moderate or severe cognitively impaired patients (i.e., Six Item Screener with three or more errors).
* Patients with Parkinson's disease (or dementia) severe enough to increase the likelihood of falling or severe enough to compromise rehabilitation.
* Likely problems, in the judgment of the investigators, with maintaining follow-up. We will, for example, exclude patients with no fixed address, those who report a plan to move out of town in the next year, or intellectually challenged patients without adequate family support.
* If the attending surgeon believes that a patient should be excluded from REGAIN because the patient is enrolled in another ongoing drug or surgical intervention trial.
* If the attending surgeon believes that there is another reason to exclude this patient from REGAIN. This reason will be documented on the case report forms.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2007-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
Rates of revision surgery | 1 year
  Revision surgery is classified as any unplanned surgery done to promote fracture healing, relieve pain, treat infection, or improve function include the following: 1) implant removal prior to fracture healing (to achieve union); 2) revision surgery with another internal fixation implant; 3) revision surgery to arthroplasty; 4) incision and drainage for deep infection at the bone implant interface; 5) correction of malunion; and 6) repair of a femoral shaft fracture.

SECONDARY OUTCOMES:
Health Related Quality of Life | Up to12 months
  HRQL will be measured using using self-administered and interview-administered questionnaires. Functional outcome questionnaires will include a generic health status measurement instrument (SF-12v2), a hip function and pain questionnaire (WOMAC), a generic utility measure (EQ-5D), the Merle d'Aubigne (MDA) pain and function score, and the Parker mobility score.
Fracture healing rates | Up to12 months
  A fracture is to be considered healed when there is obliteration of the fracture lines by newly formed bone along the cortices and within the trabecular bone on anteroposterior and lateral (or oblique) radiographs.
Complications | Up to12 months
  Complications include mortality, femoral shaft fracture, avascular necrosis, nonunion, malunion (shortening, varus deformity, valgus deformity and rotational malunion), implant breakage or failure, and infection (i.e., superficial and deep).

CONTACTS AND LOCATIONS:
Overall Officials: Mohit Bhandari, MD FRCSC MSc, Principal Investigator — McMaster University
Locations (5):
- Canada (3):
  - Hamilton General Hospital, Hamilton, Ontario
  - St. Joseph's Hospital, Hamilton, Ontario
  - St. Michael's Hospital, Toronto, Ontario
- Aarhus University Hospital, Aarhus, Denmark
- Sahlgrenska University Hospital, Gothenburg, Sweden

REFERENCES:
- [Background] Parker MJ, Pryor GA. Gamma versus DHS nailing for extracapsular femoral fractures. Meta-analysis of ten randomised trials. Int Orthop. 1996;20(3):163-8. doi: 10.1007/s002640050055. PMID 8832319
- [Background] Ahrengart L, Tornkvist H, Fornander P, Thorngren KG, Pasanen L, Wahlstrom P, Honkonen S, Lindgren U. A randomized study of the compression hip screw and Gamma nail in 426 fractures. Clin Orthop Relat Res. 2002 Aug;(401):209-22. doi: 10.1097/00003086-200208000-00024. PMID 12151898
- [Background] Harrington P, Nihal A, Singhania AK, Howell FR. Intramedullary hip screw versus sliding hip screw for unstable intertrochanteric femoral fractures in the elderly. Injury. 2002 Jan;33(1):23-8. doi: 10.1016/s0020-1383(01)00106-1. PMID 11879828